CLINICAL TRIAL: NCT01852344
Title: Behavioral Differences in Effortful Control
Acronym: BDEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chandra Sekhar Sripada, Assistant Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: K23AA020297 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-13 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Methylphenidate; Effortful Control; Attention Control; Cognitive functions
MeSH Terms: interventions — Methylphenidate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Easy (Other): Healthy participant to be given 20 mgs of a placebo one hour before task performance and will perform an easy task.
  Interventions: Drug: Placebo; Behavioral: Easy Behavioral Task
- Placebo Hard (Other): Healthy participants are given 20 mgs of placebo one hour before task performance and will perform a hard task.
  Interventions: Drug: Placebo; Behavioral: Hard Behavioral Task
- Methylphenidate Easy (Other): Healthy participants are given 20 mgs of methylphenidate one hour before task performance and will perform an easy task.
  Interventions: Drug: Methylphenidate; Behavioral: Easy Behavioral Task
- Methylphenidate Hard (Other): Healthy participants are given 20 mgs of methylphenidate one hour before task performance and will perform a hard task.
  Interventions: Drug: Methylphenidate; Behavioral: Hard Behavioral Task

INTERVENTIONS:
Drug: Methylphenidate — 20 mgs of methylphenidate or placebo to be administered one hour before task performance
  Other Names: Ritalin
  Arms: Methylphenidate Easy; Methylphenidate Hard
Drug: Placebo — 20 mgs of methylphenidate or a placebo to be administered one hour before task performance
  Other Names: sugar pill
  Arms: Placebo Easy; Placebo Hard
Behavioral: Easy Behavioral Task — Subjects do an easy version of the Letter E Task.
  Arms: Methylphenidate Easy; Placebo Easy
Behavioral: Hard Behavioral Task — Subjects do a hard version of the Letter E Task.
  Arms: Methylphenidate Hard; Placebo Hard

SUMMARY:
Effortful control refers to the mental processes that help a person to regulate his or her own attention, thoughts, and emotions. This study will examine behavioral differences in healthy individuals when performing a task that induces fatigue.

The purpose of this study is to examine the effects of methylphenidate on the cognitive functions in healthy individuals when performing fatiguing cognitive tasks.

DETAILED DESCRIPTION:
Based on the multi-source interference task, all subjects' cognitive functions will be assessed based on reaction time, reaction variability, and accuracy of performance on the attention control task.

This study aims to recruit 120 total healthy participants. Overall Safety Plan Subject Protections and Safety Monitoring

1. Confidentiality of records is assured by assigning the subjects research numbers and storing computer files without reference to name, except for a single linking file that links subject's names with their research numbers. Paper records are kept in locked file drawers in a locked room, to which only authorized research personnel have access. When the study is completed, the linking file that links subject's names with their research numbers will be permanently destroyed.
2. Furthermore, upon the event of a subject's participation being terminated, all information collected prior to the subject being removed from the study, will be destroyed.
3. Personnel involved in the study are acutely sensitive to people's unease about revealing personal information. Research personnel also take the required Program for Education and Evaluation in Responsible Research and Scholarship certification, and take the utmost precautions about protecting confidentiality. When potential subject voices their lack of interest in participating, all identifying information is destroyed. During the study, subjects are reminded that they do not have to answer questions that make them feel uncomfortable

i. Data Safety and Monitoring Plan

1. No subjects will be recruited or run until the protocol receives full review and approval by the Medical IRB at the University of Michigan. A clinical research associate will accompany all subjects throughout the study. Any minor anxiety arising during the course of the procedures will be immediately assessed, and typically managed with reassurance and simple relaxation techniques. Assessment will always include an evaluation of the subject's ability to continue in the protocol.
2. All subjects will be fully informed of all the possible side-effects that could be encountered during the study. Every measure will be taken to protect subjects against even the rarest possible side effects. Principal Investigator, Dr. Chandra Sripada, has extensive prior experience with methylphenidate and the challenges utilized in this study.
3. Subjects will be encouraged to contact the investigator if they notice any symptoms or untoward side effects. All subjects will have direct access to the phone numbers and pagers of the study coordinator and the responsible physician (Dr. Sripada), as well as a 24-hour contact number (emergency room services). This information is included in the copy of the consent forms provided to the subjects.

ii. Reporting of adverse events

Adverse events (AEs) will be recorded and tracked for these projects. Adverse events will be reported per IRBs, FDA, and NIH guidelines. An adverse event is any experience that has taken place during the course of a research project, which, in the opinion of the investigators, was harmful to a subject participating in the research, increased the risks of harm in the research, or had an unfavorable impact on the risk/benefit ratio. Adverse events will be graded using the mild, moderate, severe terminology as defined:

* Mild - Noticeable to the subject, does not interfere with the subject's daily activities, usually does not require additional therapy, dose reduction, or discontinuation of the study.
* Moderate - Interferes with the subject's daily activities, possibly requires additional therapy, but does not require discontinuation of the study.
* Severe - Severely limits the subject's daily activities and may require discontinuation of the study. This would include all adverse events defined as "Serious" by the IRBMED.

The PI will assign attribution as definitely associated, probably associated, possibly associated, or unrelated. Adverse events will also be recorded as expected or unexpected. All Serious AEs and/or unexpected AEs will be reported to the IRB, NIH, and the FDA, within 7 days of occurrence or recognition. Fatal or life-threatening adverse events will be reported to the above institutions within 24 hours. Regular annual reviews of protocol activity and all adverse events will be submitted to the IRBs and NIH. Other less serious and expected AEs will also be reported to the above institutions with compliance to their requirements.

iii. Persons responsible Chandra Sekhar Sripada and Project Coordinator Christina Bohensky will be responsible for overseeing data integrity, safety monitoring, and reporting of adverse events. During the phone conferences and semi -annual meetings adverse events, recruitment, data quality and integrity and compliance with protocols will be discussed as well.

VI. Data Analysis Regression analysis will be utilized to assess whether the dependent measures for the tasks (accuracy, reaction time) are significantly correlated with measures of trait impulsivity derived from the Barratt Impulsivity Scale-11 questionnaire. Independent samples t-tests will be used to determine whether task performance differs due to methylphenidate versus placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-35

Exclusion Criteria:

* Pregnant or nursing (females)
* Any clinically significant medical condition
* Currently taking any medications (i.e., decongestants)
* Currently taking any psychoactive medications
* Alcohol or substance abuse (current or in the past 2 years)
* Liver or Kidney disease
* Any clinically significant personal or family history of cardiac problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06-05 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Sekhar Sripada, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Rachel Upjohn Building, East Medical Campus, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Easy: Healthy participants are given a placebo (sugar pill) one hour before task performance and complete an easy version of the Letter E task.
- Placebo Hard: Healthy participants are given a placebo (sugar pill) one hour before task performance and complete a hard version of the Letter E task.
- Methylphenidate Easy: Participants are given 20 mgs of methylphenidate one hour before task performance and complete an easy version of the Letter E task.
- Methylphenidate Hard: Healthy participants are given 20 mgs of methylphenidate one hour before task performance and complete a hard version of the Letter E task.
Period: Overall Study
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard
Started | 27 | 27 | 27 | 27
Actual Participation in First Assignment | 27 | 27 | 27 | 27
Completed | 27 | 27 | 27 | 27
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Hard; Methylphenidate Hard: Healthy participants are given 20 mgs of Methylphenidate one hour before task performance and complete a hard version of the Letter E task.
- Methylphenidate Easy: Healthy participants are given 20 mgs of Methylphenidate one hour before task performance and complete an easy version of the Letter E task.
- Total: Total of all reporting groups
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 108
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants who had more than 20% error on the Letter E task were excluded from analysis.
  Participants
    number analyzed (Participants) | 24 | 23 | 23 | 24 | 94
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 24 | 23 | 23 | 24 | 94
    >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants with greater than 20% error on the Letter E task were excluded from analysis.
  years
    number analyzed (Participants) | 24 | 23 | 23 | 24 | 94
    (all) | 28.2 (4.8) | 25.8 (2.0) | 26.9 (4.3) | 26.6 (3.4) | 26.9 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants who had greater than 20% error on the Letter E task were excluded from analysis.
  Participants
    number analyzed (Participants) | 24 | 23 | 23 | 24 | 94
    Female | 17 | 15 | 14 | 13 | 59
    Male | 7 | 8 | 9 | 11 | 35
Region of Enrollment [Count of Participants; unit: Participants] — Population: Participants with greater than 20% error on the Letter E task were excluded from analysis.
  Participants
    United States: number analyzed (Participants) | 24 | 23 | 23 | 24 | 94
    United States | 24 | 23 | 23 | 24 | 94

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time on the Multi-Source Interference Task
Description: Reaction time on the Multi-Source Interference Task is measured in milliseconds. Participants were given 200 trials and their mean reaction time was calculated.
Time Frame: 20-30 minutes for task completion
Population: Participants whose accuracy on task one fell below 80% or who were greater than two standard deviation outliers in reaction time were excluded from analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard
Number analyzed (Participants) | 24 | 23 | 23 | 24
milliseconds | 300 (70) | 330 (90) | 310 (80) | 280 (70)
Statistical Analysis 1: Comparison: Placebo Easy vs Placebo Hard; Test type: Superiority; p = 0.159, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Easy vs Placebo Hard vs Methylphenidate Easy vs Methylphenidate Hard; Test type: Superiority; p = 0.159, t-test, 2 sided

2. Secondary Outcome: Accuracy on the Multi-Source Interference Task.
Description: Patients completed 200 trials and the percentage of answers correct was calculated.
Time Frame: 20-30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of answers which were correct
Groups:
- Placebo Easy: Healthy participants are given a placebo (sugar pill) one hour before task performance and complete and easy version of the Letter E task.
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard
Number analyzed (Participants) | 24 | 23 | 23 | 24
percentage of answers which were correct | 94.1 (3.5) | 94.3 (5.3) | 96.1 (3.2) | 96.6 (3.2)
Statistical Analysis 1: Comparison: Placebo Hard vs Methylphenidate Hard; Test type: Superiority; p = 0.236, t-test, 2 sided

3. Secondary Outcome: Reaction Time Variability on the Multi-Source Interference Task.
Description: Reaction time variability on the Multi-Source Interference task is defined as the number of milliseconds between an individual's lowest and highest reaction time. This is averaged across all participants.
Time Frame: 20-30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard
Number analyzed (Participants) | 24 | 23 | 23 | 24
milliseconds | 270 (50) | 320 (70) | 270 (70) | 260 (40)
Statistical Analysis 1: Comparison: Placebo Hard vs Methylphenidate Hard; Test type: Superiority; p = 0.032, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Placebo Easy | Placebo Hard | Methylphenidate Easy | Methylphenidate Hard
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes